CLINICAL TRIAL: NCT02172820
Title: Increasing Cardiac Rehabilitation Participation Among Medicaid Enrollees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Diann Gaalema, Assistant Professor of Psychiatry, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRINCN9874; P20GM103644 (NIH)
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Results first posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: Coronary Artery Disease
Keywords: cardiac rehabilitation; contingency management
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Financial incentives (Experimental): Participants receive financial incentives for completing exercise sessions.
  Interventions: Behavioral: Financial incentives
- Control (No Intervention): Participants receive an equal amount of clinical contact but no financial incentives for completing exercise visits.

INTERVENTIONS:
Behavioral: Financial incentives — Patients in the experimental group will receive financial incentives for completing exercise sessions.
  Arms: Financial incentives

SUMMARY:
Participation in outpatient cardiac rehabilitation (CR) decreases morbidity and mortality for patients hospitalized with myocardial infarction, coronary bypass surgery or percutaneous revascularization. Unfortunately, only 10-35% of patients for whom CR is indicated choose to participate. Medicaid coverage and similar state-supported insurance are robust predictors of CR non-participation. There is growing recognition of the need to increase CR among patients with this form of insurance and other economically disadvantaged patients, but there are no evidence-based interventions available for doing so. In the present study we are examining the efficacy of using financial incentives for increasing CR participation among Medicaid patients. Financial incentives have been highly effective in altering other health behaviors among disadvantaged populations (e.g., smoking during pregnancy, weight loss). For this study are randomizing 130 CR-eligible Medicaid enrollees to a treatment condition where they receive financial incentives contingent on initiation of and continued attendance at CR sessions or to a "usual-care" condition where they will not receive these incentives. Treatment conditions will be compared on attendance at CR and end-of-intervention improvements in fitness, decision making and health-related quality of life. Cost effectiveness of the treatment conditions will also be examined by comparing the costs of the incentive intervention and usual care conditions with their effects on increasing CR initiation and adherence. Should this intervention be efficacious and cost-effective, it has the potential to substantially increase CR participation and significantly improve health outcomes among low-income cardiac patients.

ELIGIBILITY:
Inclusion Criteria:

* A recent myocardial infarction, percutaneous coronary intervention, coronary artery bypass graft, heart valve replacement or repair, or stable heart failure.
* Enrolled in a state-supported insurance plan for low income individuals
* Lives in and plans to remain in the greater Burlington, Vermont area (Chittenden County) for the next 12 mos.

Exclusion criteria:

* Dementia (MMSE<20) or current untreated Axis 1 psychiatric disorder other than nicotine dependence as determined by medical history
* Non-English speaking
* Prior participation in cardiac rehabilitation
* Advanced cancer, advanced frailty, or other longevity-limiting systemic disease that would preclude CR participation
* Rest angina or very low threshold angina (<2 METS) until adequate therapy is instituted
* Severe life threatening ventricular arrhythmias unless adequately controlled (e.g. intracardiac defibrillator)
* Class 4 chronic heart failure (symptoms at rest)
* Exercise-limiting non-cardiac disease such as severe arthritis, past stroke, severe lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont, Burlington, Vermont, United States

REFERENCES:
- [Derived] Gaalema DE, Elliott RJ, Savage PD, Rengo JL, Cutler AY, Pericot-Valverde I, Priest JS, Shepard DS, Higgins ST, Ades PA. Financial Incentives to Increase Cardiac Rehabilitation Participation Among Low-Socioeconomic Status Patients: A Randomized Clinical Trial. JACC Heart Fail. 2019 Jul;7(7):537-546. doi: 10.1016/j.jchf.2018.12.008. Epub 2019 May 8. PMID 31078475

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Financial Incentives | Control
Started | 65 | 65
Completed | 65 | 65
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Financial Incentives | Control | Total
Number analyzed (Participants) | 65 | 65 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (11.0) | 55.8 (9.2) | 57.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 21 | 49
  Male | 37 | 44 | 81
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 2 | 3
  White | 62 | 61 | 123
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 65 | 65 | 130

OUTCOME MEASURES:

1. Primary Outcome: Attendance at Cardiac Rehabilitation Exercise Sessions
Description: The number of patients who completed cardiac rehabilitation (CR) as defined as greater than or equal to 30 sessions. Must have been completed within 4 months of the entry stress test.
Time Frame: Within 4 months of initial stress test
Measure: Count of Participants; unit: Participants
Arm/Group | Financial Incentives | Control
Number analyzed (Participants) | 65 | 65
Participants | 36 | 19

2. Secondary Outcome: Change in Physical Health
Description: Secondary outcomes included changes between baseline and 4-month assessment in fitness (peak oxygen uptake directly measured by expired gas analysis or estimated by metabolic equivalents), body composition (body mass index, waist circumference), and quality of life (MacNew).The MacNew was designed to evaluate how daily activities and physical,emotional and social functioning are affected by heart disease and its treatment. It consists of 27 questions grouped into 3 domains: physical, mental and social functioning. Both subscales and summary score are interpreted as scores between 1 and 7; higher scores are better, and a change of at least 0.5 is a useful indicator of the minimal important difference.Changes over time were assessed using paired differences in scores from intake to four months. Due to non-normal distributions, Wilcoxon Signed Rank Test was used. Contributions of other variables to changes in secondary outcomes were examined using analyses of covariance.
Time Frame: Intake, 4 months
Population: Despite having 65 subjects in each of the two groups (financial incentives and control), only 55 and 57 subjects were analyzed respectively. Not every subject completed the initial intake (lost contact with 10 and 8 subjects, respectively).
Measure: Mean (Full Range); unit: percentage of change
Arm/Group | Financial Incentives | Control
Number analyzed (Participants) | 55 | 57
percentage of change
  % change BMI | 0.53 [-1.35 to 1.25] | 1.87 [-1.52 to 2.06]
  % change VO2 | 6.33 [3.68 to 12.30] | 12.54 [6.01 to 21.10]
  % change Waist | -1.12 [-3.02 to 0.67] | -0.23 [-2.32 to 1.61]
  % change cardiac-specific quality of life (MacNew) | 6.63 [3.70 to 14.53] | 10.73 [6.68 to 18.35]

3. Secondary Outcome: Changes in Mental Health/Cognition
Description: The Achenbach System of Empirically Based Assessment (ASEABA) is an integrated system of multi-informant assessments, including self-reports, to measure adaptive functioning and problems. The problem items have been factor-analytically reduced to 8 syndrome scales that are consistent across age, informant and culture. Higher scores represent higher symptoms (e.g. emotional/behavioral problems). The Stop Signal Reaction Time (SSRT) task measures the ability to inhibit incorrect responses. Lower scores represent a better ability to inhibit reactions. The BRIEF-A is a rating scale developed to look at everyday behaviors associated with specific domains of executive functions in adults ages 18-90.T-scores (standardized scores) are used to interpret the individual's level of executive functioning (EF). Higher scores represent more self-reported problems. A score of 50 represents the mean.A difference of 10 from the mean indicates a difference of one standard deviation (SD).
Time Frame: Changes in socio-cognitive measures will be measures from intake to completion of intervention (4 months)
Measure: Mean (Full Range); unit: percentage of change
Arm/Group | Financial Incentives | Control
Number analyzed (Participants) | 65 | 65
percentage of change
  % change ASEABA | -2.03 [-6.68 to -0.31] | 1.03 [-1.72 to 6.10]
  % change SSRT | 3.03 [-4.87 to 25.25] | 16.10 [-1.17 to 36.78]
  % change BRIEF - A | -6.23 [-11.27 to -3.57] | 0.97 [-3.62 to 8.96]

4. Other Pre Specified Outcome: Maintenance of Physical Health Gains Following Intervention.
Description: Changes in measures of physical health and fitness (peak oxygen uptake, metabolic equivalents, waist circumference, BMI, treadmill time, smoking status, perceived quality of life) will be measured from completion of intervention (4 months) to 8 months later (1 year follow-up).
Time Frame: 4 months and 1 year.
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Maintenance of Mental Health/Cognition Scores Following Intervention.
Description: Changes in measures of mental health (Beck Depression Inventory, Adult Self-Report) as well as changes in measures of executive function (Trail Making and Tower tasks, Delay Discounting, Time Perspective Questionnaire, Stop Signal Task, Behavior Rating Inventory of Executive Function) will be measured from completion of intervention (4 months) to 8 months later (1 year follow-up).
Time Frame: 4 months and 1 year.
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Health Care Costs
Description: Health care costs (cost of delivering care at the cardiac rehabilitation clinic as well as hospital costs) will be calculated from study entry to one year follow-up.
Time Frame: From intake to one year follow-up
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Costs of Attending Care
Description: Costs to the patient of attending care (transportation, child/elder care, missed wages) will be calculated from study entry to one year follow-up.
Time Frame: Intake to 1 year follow-up
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Description: Emergency Department (ED) visits and hospitalizations were pulled from the medical record
Groups:
- Financial Incentives: Participants receive financial incentives for completing exercise sessions.
  Financial incentives: Patients in the experimental group will receive financial incentives for completing exercise sessions.
  39% fewer hospital contacts in the incentive condition (p=0.079)
Arm/Group | Financial Incentives | Control
All-Cause Mortality (participants affected / at risk) | 1/65 | 2/65
Serious Adverse Events (participants affected / at risk) | 26/65 | 27/65
Other Adverse Events (participants affected / at risk) | 25/65 | 30/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Financial Incentives (N=65) | Control (N=65)
Hospitalizations (Cardiac disorders) | 19 (28) | 18 (32)
Hospitalizations (Gastrointestinal disorders) | 3 (4) | 5 (8)
Hospitalizations (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Hospitalizations (Vascular disorders) | 2 (2) | 2 (2)
Hospitalizations (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Hospitalizations (Infections and infestations) | 2 (2) | 3 (3)
Hospitalizations (Eye disorders) | 1 (2) | 0 (0)
Hospitalizations (Renal and urinary disorders) | 1 (2) | 2 (2)
Hospitalizations (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (6)
Hospitalizations (Endocrine disorders) | 1 (1) | 1 (1)
Hospitalizations (Nervous system disorders) | 0 (0) | 3 (4)
Hospitalizations (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hospitalizations (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Financial Incentives (N=65) | Control (N=65)
Emergency Department Visit (Cardiac disorders) | 7 (7) | 18 (33)
Emergency Department Visit (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 6 (9)
Emergency Department Visit (Gastrointestinal disorders) | 4 (4) | 1 (1)
Emergency Department Visit (Blood and lymphatic system disorders) | 2 (5) | 0 (0)
Emergency Department Visit (Renal and urinary disorders) | 0 (0) | 2 (2)
Emergency Department Visit (Eye disorders) | 0 (0) | 1 (1)
Emergency Department Visit (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Emergency Department Visit (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Emergency Department Visit (Endocrine disorders) | 0 (0) | 1 (1)
Emergency Department Visit (Nervous system disorders) | 3 (4) | 4 (6)
Emergency Department Visit (Infections and infestations) | 3 (3) | 3 (3)
Emergency Department Visit (General disorders) | 7 (9) | 6 (13)
Emergency Department Visit (Musculoskeletal and connective tissue disorders) | 8 (8) | 8 (12)
Emergency Department Visit (Psychiatric disorders) | 1 (1) | 1 (1)
Emergency Department Visit (Surgical and medical procedures) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Racially homogenous patient population; Baseline assessments were conducted on site; Clinical staff could not be fully blinded; Hospitalizations outside University of Vermont Medical Center may have been missed; Small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2011-06-27): https://cdn.clinicaltrials.gov/large-docs/20/NCT02172820/Prot_000.pdf
  • Informed Consent Form (2015-03-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT02172820/ICF_001.pdf
  • Statistical Analysis Plan (2011-06-27): https://cdn.clinicaltrials.gov/large-docs/20/NCT02172820/SAP_002.pdf